CLINICAL TRIAL: NCT07004127
Title: Pneumocystis in Non-HIV Patients Over 75 Years Old: Epidemiological, Diagnostic, Microbiological and Therapeutic Characteristics
Brief Title: Pneumocystis in Patients Over 75 Year
Acronym: C_PAPY
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB_22.01.05
Record Dates: First submitted 2022-08-31; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2023-04

CONDITIONS: Pneumocystis
MeSH Terms: conditions — Pneumonia, Pneumocystis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- geriatric patient with pneumocystis: geriatric patient with pneumocystis, not HIV positive,

SUMMARY:
Pneumocystis pneumonia is an infectious disease caused by Pneumocystis jirovecii that affects the lung parenchyma preferentially. Historically described in an immunocompromised population through HIV.

Worldwide, the profile of patients affected by this pathology is changing due to two main factors:

* The sustainable stabilization of HIV patients.
* The emergence of new risk factors of immunosuppression. The geriatric population is particularly affected by these risk factors, increasing the incidence of pneumocystis in this population, which does not have HIV (solid cancer, hemopathy, immunosuppressive treatments, etc.).

There is currently no work specifically studying pneumocystis in this age group. The main objective of this study is to describe the clinical, biological and therapeutic data of a cohort of geriatric patients with pneumocystis, not carrying HIV, from January 1, 2010 to December 31, 2021, in all the centers surveyed.

ELIGIBILITY:
Inclusion Criteria

1. Patient > or equal to 75 years of age
2. Microbiological diagnosis:

   * Direct examination with standard stain, finding trophozoite and/or P.jirovecii cyst (BAL or induced sputum) And/or
   * Direct examination with immunofluorescence, finding trophozoite and/or P.jirovecii cyst (BAL or induced sputum)
   * And/or
   * Positive PCR (BAL, sputum, nasopharyngeal swab or blood) and CT < 35
3. Absence of HIV infection
4. Hospitalization in French hospitals between 2010 and 2021

Non-inclusion criteria

1. Opposition of the patient to participate to the study

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: geriatric patient with pneumocystis, not HIV positive, over 75 years old
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical data | From DAY 0 to end of treatment
  description of clinical data
Therapeutic data | From DAY 0 to end of treatment
  description of treatment provide to treat pneumocystosis
Biological data | From DAY 0 to end of treatment
  Analysis of biological data realized during follow up

CONTACTS AND LOCATIONS:
Overall Officials: Adrien BARRAUD, Principal Investigator — CHU NIMES; Albert SOTTO, Md, PhD, Study Director — CHU NIMES
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: No